CLINICAL TRIAL: NCT00763191
Title: Analysis of Oculo-motor Deficiencies Associated With FMR1 Gene Expression (Genetic Abnormality Predisposing to a Neurodegenerative Disease)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: departure of the principal investigator and nobody else was able to continue this study.
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 07/10-Z
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Pre-mutation on FMR1 Gene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: examination of ocular movements
Other: MATTIS test
Other: UPDRS test
Other: CRST test

SUMMARY:
The specific aim of this study is to compare ocular movements abnormalities between males with pre-mutation on FRM1 gene (symptomatic or asymptomatic on the motor plan and/or on the cognitive plan), males without the pre-mutation and males with multi-systematized atrophy, in order to identify the neuronal structures implicated in this pathology.

DETAILED DESCRIPTION:
Patient will be followed at the Nantes hospital during half a day for :

* examination of ocular movements
* performing Neuro-psychological test (MATTIS)
* performing tests with scales of motricity (UPDRS, CRST, ICARS).

ELIGIBILITY:
FOR PATIENTS WITH PREMUTATION ON FMR1 GENE (30 patients expected):

Inclusion criteria:

* Male
* > or equal to 50 years old
* Ally second or third degree with a child affected of "fragile X"
* Not living far from Nantes so that visits to the Nantes hospital can be easy
* Pre-mutation on FMR1 gene
* Signed informed consent

Exclusion criteria:

* Female
* <50 years old
* visual acuteness < 1/10
* MATTIS dementia scale <100 (normal:144)
* Occurrence, shown by MRI (Magnetic Resonance Imaging), of a pathology either ischemic vascular or hemorrhagic or tumoral

FOR PATIENTS WITHOUT PRE-MUTATION ON FMR1 GENE (10 patients expected):

Inclusion criteria:

* Male
* > or equal to 50 years old
* Ally second or third degree with a child affected of "fragile X"
* Not living far from Nantes so that visits to the Nantes hospital can be easy - Signed informed consent

Exclusion criteria:

* Female
* <50 years old
* visual acuteness < 1/10
* MATTIS dementia scale <100 (normal:144)
* Pre-mutation on FMR1 gene
* Occurrence, shown by MRI, of a pathology either ischemic vascular or hemorrhagic or tumoral

FOR PATIENTS WITH MULTI-SYSTEMATIZED ATROPHY (10 patients expected):

Inclusion criteria:

* Male
* > or equal to 50 years old
* Not living far from Nantes so that visits to the Nantes hospital can be easy
* "probable" diagnosis of multi-systematized atrophy
* Signed informed consent

Exclusion Criteria:

* Female
* <50 years old
* visual acuteness < 1/10
* MATTIS dementia scale <100 (normal:144)
* Occurrence, shown by MRI, of a pathology either ischemic vascular or hemorrhagic or tumoral

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Comparison of the oculo-motricity of patients with FMR1 pre-mutation with the oculo-motricity of patients without FMR1 pre-mutation

SECONDARY OUTCOMES:
Comparison of the oculo-motricity of patients with FMR1 pre-mutation with the oculo-motricity of patients with multi-systematized atrophy
Analysis of the correlation between the genotype (number of CGG repetition) and the phenotype.
For subjects with FMR1 pre-mutation, comparison of the neuro-psychological test results to the oculo-motor abnormalities.

CONTACTS AND LOCATIONS:
Locations (1):
- Laennec hospital, university hospital of Nantes, Nantes, France